CLINICAL TRIAL: NCT05966688
Title: A Phase 1 Study to Evaluate the Effect of Co-administration on the Pharmacokinetics of SPR720, Azithromycin, and Ethambutol in Healthy Volunteers
Brief Title: A Study to Evaluate the Effect of Co-administration on the Pharmacokinetics of SPR720, Azithromycin, and Ethambutol in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPR720-102
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Azithromycin; Ethambutol

STUDY DESIGN:
Intervention Model Description: It is anticipated that participants will enroll one after another in each arm of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- SPR720 1000 mg (Experimental): Healthy participants will receive SPR720 1000 milligrams (mg), orally, once daily (QD) for 7 days.
  Interventions: Drug: SPR720
- Azithromycin 500 mg (Experimental): Healthy participants will receive azithromycin 500 mg, orally, QD for 7 days.
  Interventions: Drug: Azithromycin
- Ethambutol 800 mg (Experimental): Healthy participants will receive ethambutol 800 mg, orally, QD for 7 days.
  Interventions: Drug: Ethambutol
- SPR720 1000 mg + Azithromycin 500 mg + Ethambutol 800 mg (Experimental): Healthy participants will be co-administered SPR720 1000 mg, azithromycin 500 mg, and ethambutol 800 mg, orally, QD for 7 days.
  Interventions: Drug: SPR720; Drug: Azithromycin; Drug: Ethambutol
- Azithromycin 500 mg + Ethambutol 800 mg (Experimental): Healthy participants will be co-administered azithromycin 500 mg, and ethambutol 800 mg, orally, QD for 7 days.
  Interventions: Drug: Azithromycin; Drug: Ethambutol

INTERVENTIONS:
Drug: SPR720 — Multiple oral doses of SPR720 capsules.
  Arms: SPR720 1000 mg; SPR720 1000 mg + Azithromycin 500 mg + Ethambutol 800 mg
Drug: Azithromycin — Multiple oral doses of azithromycin.
  Arms: Azithromycin 500 mg; Azithromycin 500 mg + Ethambutol 800 mg; SPR720 1000 mg + Azithromycin 500 mg + Ethambutol 800 mg
Drug: Ethambutol — Multiple oral doses of ethambutol.
  Arms: Azithromycin 500 mg + Ethambutol 800 mg; Ethambutol 800 mg; SPR720 1000 mg + Azithromycin 500 mg + Ethambutol 800 mg

SUMMARY:
The primary purpose of this study is to evaluate the pharmacokinetics (PK) of SPR720, azithromycin, and ethambutol, administered separately and co-administered, in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between ≥18.0 and ≤32.0 kilograms per meter square (kg/m^2) and weight between 50.0 and 100.0 kilograms (kg) (inclusive) at the Screening visit.
* Medically healthy without clinically significant medical history, abnormalities in physical examination, laboratory tests, vital signs, or electrocardiogram (ECG) at the Screening visit.
* Has suitable venous access for repeated blood sampling.
* Has ability and willingness to abstain from alcohol, caffeine, xanthine-containing beverages or food (coffee, tea, chocolate, and caffeine-containing sodas, colas, etc.) or products containing any of these from 48 hours prior to study drug administration until discharge from the clinical research unit (CRU).

Exclusion Criteria:

* Has a history of clinically significant acute illness or surgery within the previous 3 months prior to Screening Visit or Day -1.
* Has a known history of clinically significant hypersensitivity reaction or anaphylaxis to any medication.
* Has any condition possibly affecting drug absorption (e.g., previous surgery on the gastrointestinal tract [including removal of parts of the stomach, bowel, liver, gall bladder, or pancreas]). History of uncomplicated appendectomy ≥1 year prior to Screening Visit would not be considered exclusionary at the discretion of the Investigator.
* Is unable to swallow the dosage forms.
* Has received any other investigational medicinal product or participation in another investigational clinical study that included drug treatment within 30 days prior to Day 1 dose (based on the timing of the last Follow-up Visit for the previous study to Day 1 of the current study).

[Note: Other inclusion and exclusion criteria as per protocol may apply.]

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Study Drug | Pre-dose and at multiple time points post-dose up to Day 8
Time to Attain Maximum Plasma Concentration (tmax) for Study Drug | Pre-dose and at multiple time points post-dose up to Day 8
Area Under the Concentration-time Curve From Time Zero to Dosing Interval (AUC0-τ) for Study Drug | Pre-dose and at multiple time points post-dose up to Day 8

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | From the first dose of study drug through follow-up Day 13

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No